CLINICAL TRIAL: NCT06081179
Title: Does Serotonin System Stimulation Increase Pro-social Behavior? - A Comparative Pharmacological Neuroscientific Study in Healthy Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2A-SC-1
Record Dates: First submitted 2023-09-25; First posted 2023-10-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: MDMA; Psilocybin; Methylphenidate; pro-social behavior; healthy controls; psychedelics; serotonin
MeSH Terms: interventions — Psilocybin; N-Methyl-3,4-methylenedioxyamphetamine; Methylphenidate

STUDY DESIGN:
Intervention Model Description: single-center, double-blind, parallel-group, randomized study design
Who Masked: Participant, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Psilocybin (Active Comparator): 40 participants will receive psilocybin
  Interventions: Drug: Psilocybin
- MDMA (Active Comparator): 40 participants will receive MDMA
  Interventions: Drug: 3,4 Methylenedioxymethamphetamine
- Methylphenidate (Active Comparator): 40 participants will receive methylphenidate
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Psilocybin — Single dose of psilocybin (15mg), orally in form of capsules
  Other Names: magic mushrooms
  Arms: Psilocybin
Drug: 3,4 Methylenedioxymethamphetamine — Single dose of MDMA (100mg), orally in form of capsules
  Other Names: MDMA; Ecstasy
  Arms: MDMA
Drug: Methylphenidate — Single dose of methylphenidate (60mg), orally in form of capsules
  Other Names: Ritalin
  Arms: Methylphenidate

SUMMARY:
The study looks into whether administering psychedelic substances that stimulate the serotonin system influences pro-social behavior when compared to administering substances that stimulate the dopamine system in healthy individuals.

DETAILED DESCRIPTION:
Psychedelic substances have been shown to be powerful modulators of social perception and behavior during the acute experience. This is of particular interest given that social relationships play a key role in the development and resolution of psychiatric symptoms. However, the neuropharmacological mechanism underlying pro-social effects and time-dependent changes currently remain unclear. This study therefore aims at answering two key questions: 1) Does stimulation of the serotonin system induce lasting effects on pro-social behavior? and 2) Are these effects specific to serotonergic stimulation? The following proposed study will assess these questions by investigating objective, ecologically valid measures of pro-social cognition four weeks after different pharmacological challenges (MDMA, an entactogen and releaser of serotonin, norepinephrine, and dopamine; psilocybin: a classical psychedelic and serotonin 2A receptor agonist, methylphenidate: an amphetamine and norepinephrine-dopamine re-uptake inhibitor) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female at the age of 18-40
* Willing and capable to give informed consent for study participation as documented by signature (Informed Consent Form) after the nature of the study has been thoroughly explained
* Willing to refrain from drinking alcohol the day before testing session, from drinking alcohol and caffeinated drinks at the testing days and from consuming psychoactive substances two weeks before the first investigation visit and for the duration of the study
* Willing to abstain from using drugs that may interfere with the effects of the study medications including sleeping aids, cough medications, beta-blocker or other substances with potentially relevant psychoactive and cardiovascular effects.
* Able and willing to comply with all study requirements
* Good physical health with no unstable medical conditions, as determined by medical history, physical examination, routine blood labs, electrocardiogram, urine analysis, and urine toxicology
* Women of childbearing potential (as defined by: 'the age of carrying or giving birth to a child', normally between 14-45 years of age, not in menopause, last menstrual period (LMP) less than 12 months, no removal of ovaries or uterus, no ligature of Fallopian tubes') must be using an effective, established method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices. Note: female participants who are surgically sterilized/hysterectomized or post-menopausal for longer than 2 years are not considered as being of childbearing potential
* Willing not to drive a traffic vehicle or to operate machines within 48h following substance administration
* Have a family member or friend who can pick them up after the substance administration sessions (driving is forbidden at drug treatment days)

Exclusion Criteria:

* Poor knowledge of the German language
* Previous significant adverse response to a hallucinogenic drug (incl. psilocybin), MDMA, or methylphenidate
* Allergy or hypersensitivity to previous use of MDMA, psilocybin, or methylphenidate
* Lifetime history of hallucinogen (incl. psilocybin), MDMA, or methylphenidate use on more than 10 occasions
* Personal and family history of major psychiatric disease (e.g., schizophrenia, schizoaffective disorder, psychosis, major depression, bipolar disorder, psychotic disorder, substance addiction/abuse other than caffeine and nicotine) as defined in the DSM-V (1st and 2nd degree relatives)
* History of suicidal behavior
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia, etc. of the participant
* Attention-Deficit/Hyperactivity-Disorder (ADHD)
* Any current major medical condition (e.g., neurologic, cardiovascular, metabolic, infectious disease) or any unstable illness as determined by medical history or laboratory tests
* Uncorrected hypo-or hyperthyroidism
* Uncorrected hypo-and hypertension
* Epilepsy
* Abnormal electrocardiogram
* BMI <17 or >35
* Personal history of head trauma, brain/cardiac surgery, fainting, or electroconvulsive therapy
* Personal and family history of seizure disorder and strokes (1st and 2nd degree relatives)
* Participation in another study where pharmaceutical compounds are given within the 30 days preceding and during the present study
* Current psychopharmacological treatment or medication that affects brain function
* Use of medications that are contraindicated or otherwise interfere with the effects of the study medications (monoamine oxidase inhibitors, antidepressants, sedatives etc.)
* Women who are pregnant or breast feeding, or have the intention to become pregnant during the study (for safety reasons, a urine pregnancy test will be done at the screening visit and before the substance administration)
* Enrollment of the investigator, his/her family members, employees, and other dependent persons

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Multifaceted Empathy Test | t0 - 10 days (+/- 7 days) and t0 + 4 weeks (+/- 3 days); t0 being the day of substance administration
  The Multifaceted Empathy Test is a task assessing the cognitive and emotional aspects of empathy. Participants process 40 photos of people in emotionally charged situations. Each aspect of empathy (implicit and explicit emotional empathy, and cognitive empathy) is tested with 20 positive valence stimuli and 20 negative valence stimuli, yielding a total of 120 trials.
Moral Inference Task | t0 - 10 days (+/- 7 days) and t0 + 4 weeks (+/- 3 days); t0 being the day of substance administration
  The Moral Inference task is an approach to evaluate the computational basis of moral inference and its temporal dynamics. Participants observe and predict the decisions of two "agents" who repeatedly choose on administering painful electric shocks to another person in a different room in return for money, and rate them every third trial for their moral character. At the end of the game there is a short trust game. Participants can win actual money in this game (up to 1 CHF).
Zurich Prosocial Game | t0 - 10 days (+/- 7 days) and t0 + 4 weeks (+/- 3 days); t0 being the day of substance administration
  The Zurich Prosocial Game is a computer-based pro-social game which allows for assessment of prosocial behavior, considering the influence of helping cost, distress cues in helping behavior, and reciprocity on pro-social behavior through different trial types. Participants can win actual money in this game (up to 6.50 CHF).
Social Gaze Task | t0 - 10 days (+/- 7 days) and t0 + 4 weeks (+/- 3 days); t0 being the day of substance administration
  The Social Gaze Task is a paradigm in which participants' gaze is used to control the gaze of a tropomorphic virtual figure. The aim is to capture the reciprocal and interactive nature of joint attention. Participants' gaze behavior is recorded using an eye-tracking device. The outcome measures we will use are pupil size, valence, and arousal ratings.
Moral Expansion Task | t0 - 10 days (+/- 7 days) and t0 + 4 weeks (+/- 3 days); t0 being the day of substance administration
  In the Moral Expansion Task, the influence of social distance is elicited by having participants indicate countries with different social distances and decide how much money out of CHF 100 they would like to donate to the Red Cross in each country. One participant's choice is then randomly selected, and the donation is implemented while the chosen participant receives the remaining amount.
Social Network Questionnaire | t0 - 10 days (+/- 7 days) and t0 + 4 weeks (+/- 3 days); t0 being the day of substance administration
  The Social Network Questionnaire is used to assess the size of a person's social network and the emotional support and strain experienced from that network. Participants provide the initials of personal contacts from various domains with whom they have had contact with in the past 4 weeks. 28 items are rated on a 6-point scale, asking how much emotional support and emotional burden they have felt from their social contacts. The total score for those items ranges from 28 to 168.
Pro-social Voting Behavior | t0 - 10 days (+/- 7 days) and t0 + 4 weeks (+/- 3 days); t0 being the day of substance administration
  The Pro-social Voting Behavior is used to evaluate pro-social voting behavior as a real-world measure of social behavior. The scale consists of 11 items. Each item is rated on a 4-point scale. The total score ranges from 11 to 44. Not all items are accounted equally to capture pro-social voting behavior, as some are reversed.
Oxford Utilitarianism Scale | t0 - 10 days (+/- 7 days) and t0 + 4 weeks (+/- 3 days); t0 being the day of substance administration
  The Oxford Utilitarianism Scale measures two dimensions of utilitarian tendencies. The scale consists of 9 items. Each item is rated on a 7-point scale. The total score ranges from 9 to 63.
Compassion Scale | t0 - 10 days (+/- 7 days) and t0 + 4 weeks (+/- 3 days); t0 being the day of substance administration
  The Compassion Scale measures an individual's level of compassion towards others. The scale consists of 16 items. Each item is rated on a 5-point scale. The total score ranges from 16 to 80.
Inclusion of others in the self | t0 - 10 days (+/- 7 days), t0, and t0 + 4 weeks (+/- 3 days); t0 being the day of substance administration
  The Inclusion of others in the self is designed to assess the perceived relationship between an individual's self and other people/all living things. It consists of two items. Each item is rated as circles corresponding to a numerical score, ranging from 1 to 8. The total score ranges from 2 to 16.

SECONDARY OUTCOMES:
5-Dimensional Altered States of Consciousness Rating Scale | t0 (the day of substance administration)
  The 5-Dimensional Altered States of Consciousness Rating Scale measures subjective experiences of altered states of consciousness. It contains 94 items, which are formulated as a visual analog scale, assessing different dimensions of altered states of consciousness.
5-Dimensional Altered States of Consciousness Rating Scale short | t0 (the day of substance administration)
  The 5-Dimensional Altered States of Consciousness Rating Scale short is a shorter version of the 5-Dimensional Altered States of Consciousness Rating Scale for measuring subjective experiences of altered states of consciousness. The scale consists of 15 items chosen from the full version, which are formulated as a visual analog scale.
Mystical Experience Questionnaire | t0 (the day of substance administration)
  The Mystical Experience Questionnaire is used to assess mystical experiences. The scale consists of 30 items. Each item is rated on a 6-point scale (from 0 to 5). The total score ranges from 0 to 150.
Persisting Effects Questionnaire | t0 + 4 weeks (+/- 3 days) and t0 + 16 weeks (+/- 7 days); t0 being the day of substance administration
  The Persisting Effects Questionnaire is used to assess changes in attitudes, moods, behavior, and spiritual experience. The scale consists of 144 items. 140 items are rated on a 6-point scale (from 0 to 5). The last four items use different scaling. The total score ranges from 4 to 724.
Epistemic and personal transformation (pre and post versions) | t0 (the day of substance administration)
  The Epistemic and personal transformation is used to capture the intensity and qualities of epistemic and personal transformation and participants' expectations and desires thereof. Both pre and post versions include open questions and 4 items that are rated on a visual analog scale from 0 to 100. The total score ranges from 0 to 400 for pre and post versions each. The post version additionally captures the substance intake assumption of the participants.
Symptom Checklist 90-R | t0 - 10 days (+/- 7 days) and t0 + 16 weeks (+/- 7 days); t0 being the day of substance administration
  The Symptom Checklist 90-R is used to assess a broad range of psychological problems and symptoms of psychopathology within the past seven days. It consists of 90 items. Each item is rated on a 5-point scale (from 0 to 4). The total score ranges from 0 to 360.
The Positive and Negative Affect Schedule | t0 - 10 days (+/- 7 days), t0, t0 + 4 weeks (+/- 3 days), and t0 + 16 weeks (+/- 7 days); t0 being the day of substance administration
  The Positive and Negative Affect Schedule is used to assess both positive and negative affect. It consists of two 10-item scales, one measuring positive affect and one measuring negative affect. Each item is rated on a 5-point scale (from 0 to 4). The total scores range from 0 to 80.
FEELINGS | t0 - 10 days (+/- 7 days) and t0 + 16 weeks (+/- 7 days); t0 being the day of substance administration
  The FEELINGS scales consist of a series of six short questionnaires to assess regulation, self-esteem, satisfaction with life, life orientation, and meaning in life. Emotional Regulation Questionnaire uses a 7-point scale with a total score range from 7 to 70 (10 items). Satisfaction with Life Scale uses a 7-point scale with a total score range from 5 to 35 (5 items). Rosenberg Self-Esteem Scale uses a 4-point scale with a total score range from 10 to 40 (10 items). Life Orientation Test-Revised uses a 5-point scale with a total score range from 10 to 50 (10 items). Lebenssinn-Fragebogen uses a 7-point scale with a total score range from 10 to 70 (10 items). HSF uses a 5-point scale with a total score range from 6 to 30 (6 items).
Ego Consciousness Change of Perspective Questionnaire (1 & 2) | t0 and t0 + 4 weeks (+/- 3 days); t0 being the day of substance administration
  Ego Consciousness Change of Perspective Questionnaire is used to measure the two dimensions Consciousness and Ego. Questions for the acute effects of substance intake (27 items) and questions for the longer-lasting effects (6 items) are included. Each item is rated on a visual analog scale from 0 to 100. The total score ranges from 0 to 3300.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatrische Universitätsklinik Zürich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Preller KH, Vollenweider FX. Modulation of Social Cognition via Hallucinogens and "Entactogens". Front Psychiatry. 2019 Dec 3;10:881. doi: 10.3389/fpsyt.2019.00881. eCollection 2019. PMID 31849730
- [Background] Cruwys T, Haslam SA, Dingle GA, Haslam C, Jetten J. Depression and Social Identity: An Integrative Review. Pers Soc Psychol Rev. 2014 Aug;18(3):215-238. doi: 10.1177/1088868314523839. Epub 2014 Apr 12. PMID 24727974